CLINICAL TRIAL: NCT05024214
Title: Envafolimab(KN035) in Combination With Lenvatinib in the Treatment of Advanced Solid Tumors: a Multicenter, Open-label, Phase Ib/II Study
Brief Title: Phase Ib/II Trial of Envafolimab Plus Lenvatinib for Subjects With Solid Tumors
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: 3D Medicines (Sichuan) Co., Ltd. (Industry)
Responsible Party: Sponsor
Organization: 3D Medicines (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KN035-CN-010
Record Dates: First submitted 2021-08-15; First posted 2021-08-27 (Actual); Last update posted 2025-05-29 (Actual); Status verified 2025-05

CONDITIONS: Solid Tumors; Non-small Cell Lung Cancer; Renal Cell Carcinoma; Hepatocellular Carcinoma
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Carcinoma, Renal Cell; Carcinoma, Hepatocellular | interventions — lenvatinib; envafolimab; Sunitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Phase Ib arm (Experimental): Subjects with advanced or metastatic solid tumor (excluding hepatocellular carcinoma and thyroid cancer) with disease progression or intolerance or no effective treatment after standard therapy
  Interventions: Drug: Lenvatinib + Envafolimab
- Phase II cohort1-NSCLC (Experimental): Subjects with non-small cell lung cancer, resistant after previous treatment with PD-(L)1 inhibitors
  Interventions: Drug: Lenvatinib + Envafolimab
- II Phase cohort1-RCC (Experimental): Subjects with renal cell carcinoma, resistant after previous treatment with PD-(L)1 inhibitors
  Interventions: Drug: Lenvatinib + Envafolimab
- Phase II cohort1-HCC (Experimental): Subjects with hepatocellular carcinoma, resistant after previous treatment with PD-(L)1 inhibitors
  Interventions: Drug: Lenvatinib + Envafolimab
- Phase II cohor2-experiment group (Experimental): Subjects with renal cell carcinoma, no previous systemic treatment for advanced disease
  Interventions: Drug: Lenvatinib + Envafolimab
- Phase II cohort2-control group (Experimental): Subjects with renal cell carcinoma, no previous systemic treatment for advanced disease
  Interventions: Drug: Sunitinib

INTERVENTIONS:
Drug: Lenvatinib + Envafolimab — Lenvatinib will be administered with water orally once a day (with or without food) continuously in 28-day treatment cycle.
  Envafolimab, 400 mg per dose, subcutaneous injection, dosed on D1 and then D15 of Treatment Cycle 1, and D1 of Treatment Cycle 2 and every subsequent cycles, with every 28 days as one treatment cycle.
  Arms: II Phase cohort1-RCC; Phase II cohor2-experiment group; Phase II cohort1-HCC; Phase II cohort1-NSCLC; Phase Ib arm
Drug: Sunitinib — Sunitinib will be administered with water orally once daily, on a schedule of 4 weeks on treatment followed by 2 weeks off (Schedule 4/2) in 42-day treatment cycle.
  Arms: Phase II cohort2-control group

SUMMARY:
This is an open-label, multi-center study of Phase Ib/II study to assess the efficacy and safety of Envafolimab combinded with Lenvatinib in the treatment of subjects with advanced solid tumors. The primary hypothesis of this study is that subjects will have a better objective response rate (ORR) when treated with Envafolimab plus Lenvatinib than SOC.

ELIGIBILITY:
Inclusion Criteria:

1. Eighteen years and older;
2. phase Ib:Histological or cytological diagnosis of Locally advanced or metastatic solid tumors (excluding hepatocellular carcinoma and thyroid carcinoma) that have progressed after standard treatment or are intolerant or have no effective treatment;
3. phase II cohort 1:Histological or cytological diagnosis of NSCLC，RCC, HCC, resistance to previous treatment with PD-(L)1 inhibitor; previous system treatment lines≤2;
4. phase II cohort 2：Unresectable locally advanced or metastatic or recurrent RCC;
5. Tumor tissue samples or biopsies from FFPE archived or fresh biopsies with locally advanced/metastatic disease must be provided, and if biopsies are not available, samples obtained prior to receiving adjuvant/neoadjuvant chemotherapy are allowed;
6. phase Ib and phase II cohort 1: Eastern Cooperative Oncology Group(ECOG) Performance Status of 0 or 1; Phase II cohort 2: Karnofsky physical status (KPS) assessment ≥70；
7. Life expectancy of at least 12 weeks;
8. At least one measurable lesion per RECIST 1.1;
9. Adequate organ function;
10. Signed informed consent.

Exclusion Criteria:

1. Prior anticancer treatment within 4 weeks prior to the first dose of study drugs;
2. Toxicity from prior anticancer therapy prior to the first dose of study drugs not recovered to ≤ grade1;
3. Hypertension did not satisfactory controlled after antihypertensive medication
4. Phase Ib/II: Subjects who were previously treated with Lenvatinib or who participated in a clinical trial of a generic version of Lenvatinib
5. Phase II cohort 1, intolerance to treatment with A PD-(L)1 inhibitor; History of severe digestive disease that can affect the oral absorption of Lenvatinib/Sunitinib;
6. Uncontrollable or significant cardiovascular or cerebrovascular disease;
7. Active, known history or suspected autoimmune disease;
8. Have used or require treatment with >10 mg/day of prednisone or an equivalent dose of systemic corticosteroids within 14 days prior to the first dose of study drugs;
9. have received live attenuated vaccine within 28 days prior to the first study drug treatment or are scheduled to receive it during the study period;
10. Subjects with known or suspected interstitial pneumonia;
11. Any serious active infection requiring systemic antibacterial, antifungal or antiviral therapy at screening, including active tuberculosis; Known history of human immunodeficiency virus (HIV) infection or acquired immunodeficiency syndrome (AIDS)
12. Active hepatitis B or hepatitis C;
13. Known history of severe gastrointestinal bleeding or active hemoptysis or other severe bleeding within 6 months prior to first study drug therapy;
14. Uncontrolled pleural effusion, pericardial effusion, or ascites requiring repeated drainage ;
15. Known active or symptomatic central nervous system (CNS) metastases and/or carcinomatous meningitis;
16. Have other primary malignancies within 5 years;
17. Known history of contraindications or hypersensitivity reactions to any investigational drug component or any known excipients
18. Women who are pregnant or breastfeeding.
19. Radiographic evidence of major blood vessel invasion/infiltration may be considered for enrollment if the investigator assesses that the risk is manageable.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 170 (Estimated)
Dates: Start 2021-11-15 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
RP2D(Phase Ib) | first Cycle (28 Days)
  Recommendation phase II dose
Dose Limiting Toxicity (DLT) (Phase Ib) | first Cycle (28 Days)
  Number of participants who experience DLT of the first Cycle（28days)
objective response rate (ORR) （Phase II） | Two years
  Defined as the percentage of participants in the analysis population who experienced a Complete Response or a Partial Response and was assessed using RECIST 1.1 based on investigator evaluation.

SECONDARY OUTCOMES:
Objective response rate (ORR) （Phase Ib） | Two years
  Defined as the percentage of participants in the analysis population who experienced a Complete Response or a Partial Response and was assessed using RECIST 1.1 based on investigator evaluation.
Duration of response (DoR) | Two years
  Defined as the time from response to documented disease progression per Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST 1.1) based on investigator evaluation.
Progression Free Survival (PFS) | Two years
  Defined as the time from experiment drug administration to documented disease progression per Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST 1.1) or death due to any cause, whichever occurred first and was based on investigato evaluation.
Overall Survival (OS) | Two years
  Defined as the time from experiment drug administration to death due to any cause

OTHER OUTCOMES:
Disease control rate (DCR) | Two years
  Defined as the percentage of participants in the analysis population who experienced a Complete Response or a Partial Response or stable disease and was assessed using RECIST 1.1 based on investigato evaluation
Time to Response(TTR) | Two years
  Defined as the time from experiment drug administration to the first date of response was objectively documented

CONTACTS AND LOCATIONS:
Overall Officials: Tianshu Liu, Principal Investigator — Fudan University
Locations (23):
- China (23):
  - The First Affiliated Hospital of Bengbu Medical College, Bengbu, Anhui
  - The Seventh Medical Center of the PLA General Hospital, Beijing, Beijing Municipality
  - Beijing Hospital, Beijing, Beijing Municipality
  - Fujian Medical University Union Hospital, Fuzhou, Fujian
  - Zhongshan Hospital,Fudan University(Xiamen Branch), Xiamen, Fujian
  - Dongguan People's Hospital, Dongguan, Guangdong
  - Zhujiang Hospital of Southern Medical University, Guangzhou, Guangdong
  - The Fifth Affiliated Hospital Sun Yat-Sen University, Zhuhai, Guangdong
  - Harbin Medical University Cancer Hospital, Haerbin, Heilongjiang
  - The First Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan
  - The Second Affiliater Hospital of Nanchang University, Nanchang, Jiangxi
  - THE First Hospital of Jilin University, Changchun, Jilin
  - Jilin Cancer Hospital, Changchun, Jilin
  - The First Affiliated Hospital of Dalian Medical University, Dalian, Liaoning
  - Shengjing Hospital of China Medical University, Shenyang, Liaoning
  - Liaoning Cancer Hospital & Institute, Shenyang, Liaoning
  - The 960th Hospital of the PLA Joint Logistics Support Force, Jinan, Shandong
  - First Hospital of Shanxi Medical University, Taiyuan, Shanxi
  - Tianjin Medical University Cancer Institute & Hospital, Tianjin, Tianjin Municipality
  - The Cancer Affiliated Hospital of Xinjiang Medical College, Ürümqi, Xinjiang
  - Yunnan Cancer Hospital, Kunming, Yunnan
  - Sir Run Run Shaw Hospital Zhejiang University School of Medicine, Hangzhou, Zhejiang
  - Fudan University, Shanghai

IPD SHARING:
Plan to Share IPD: Undecided